CLINICAL TRIAL: NCT07149740
Title: Data Gathering for A10900
Status: Recruiting | Type: Observational
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Other Study IDs: OPT1110
Record Dates: First submitted 2025-07-11; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Retinal Disease; Healthy; Glaucoma; Corneal Diseases
MeSH Terms: conditions — Retinal Diseases; Glaucoma; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Retinal Disease
  Interventions: Device: OCT
- Healthy
  Interventions: Device: OCT
- Glaucoma
  Interventions: Device: OCT
- Corneal Disease
  Interventions: Device: OCT

INTERVENTIONS:
Device: OCT — A10900 is an optical coherence tomography device

SUMMARY:
The objective of this study is to gather Optical Coherence Tomography (OCT) data on normal and diseased eyes

ELIGIBILITY:
Inclusion/Exclusion Criteria Inclusion Criteria for Retinal Disease Group

1. Participants 22 years of age or older on the date of informed consent
2. Participants able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. BCVA 20/400 or better in the study eye
4. Participants presenting at the site with retinal disease
5. Diagnosis of some type of retinal pathology by investigator, may include, but not limited to: Macular Degeneration (including participants with drusen and geographic atrophy and choroidal neovascularization), Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Central Serous Retinopathy and others

Exclusion Criteria for Retinal Disease Group

1. Participants unable to tolerate ophthalmic imaging
2. Participants not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Participant has a condition or is in a situation which the investigator feels may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study
4. Presence of glaucoma or any ocular pathology other than a retinal pathology in the study eye as determined by self-report and/or investigator assessment at the study visit;

Inclusion Criteria for Glaucoma Group

1. Participants 22 years of age or older on the date of informed consent
2. Participants able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. BCVA 20/40 or better in the study eye
4. History of Visual field defects within the previous year from the study visit or measured the day of the study visit consistent with glaucomatous optic nerve damage with at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."
5. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

   1. Diffuse thinning, focal narrowing, or notching of the neuroretinal rim, especially at the inferior or superior poles with or without disc hemorrhage;
   2. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue

Exclusion Criteria for Glaucoma Group

1. Participants unable to tolerate ophthalmic imaging
2. Participants not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Participant has a condition or is in a situation which the investigator feels may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study
4. No reliable visual field test result within the previous year from the study visit, defined as fixation losses > 33% or false positives > 33%, or false negatives > 33% in the study eye
5. Presence of any ocular pathology except glaucoma in the study eye Inclusion Criteria for Corneal Group

1. Participants 22 years of age or older on the date of informed consent 2. Participants able to understand the written informed consent and willing to participate as evidenced by signing the informed consent 3. Participants presenting at the site with corneal disease, for example but not limited to, corneal disorders due to contact lens wear, post-refractive surgery, dry eye, keratoconus 4. Participant is able to comply with the study procedures.

Exclusion Criteria for Corneal Group

1. Participants unable to tolerate ophthalmic imaging
2. Participant has a condition or is in a situation which the investigator feels may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study
3. Participant with ocular media not sufficiently clear to obtain acceptable OCT images.

Inclusion Criteria for Normal Group

1. Participants 22 years of age or older on the date of informed consent
2. Participants able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Participants presenting at the site with normal eyes (Cataracts, LASIK, PRK, and peripheral pathology that does not affect the posterior pole region, for example lattice and peripheral drusen, are allowed).
4. BCVA 20/40 or better (each eye)
5. Participant is able to comply with the study procedures

Exclusion Criteria for Normal Group

1. Participants unable to tolerate ophthalmic imaging
2. Participant has a condition or is in a situation which the investigator feels may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study
3. Participant with ocular media not sufficiently clear to obtain acceptable OCT images
4. History of leukemia, dementia or multiple sclerosis

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with healthy, glaucoma, retinal disease and corneal disease located in different geographic locations in the US
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of OCT Scans | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ketchum Health, Anaheim, California
  - Eye Care and Laser Surgery of Newton Wellselley, Wellesley Hills, Massachusetts
  - Charles Retina Institute, Germantown, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
This is included in the participant's informed consent. Images, demographics, ophthalmic assessments and examinations, visual fields, and ophthalmic and medical history.